CLINICAL TRIAL: NCT05317793
Title: Ambulatory Electrodermal Activity Measurements as Part of Identification and Prevention of Job Burnout
Status: Active, not recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: R21149
Record Dates: First submitted 2022-03-14; First posted 2022-04-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Burnout, Professional; Mental Health Issue; Anxiety; Depression
MeSH Terms: conditions — Burnout, Professional; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Professionals: 150 knowledge workers from three Finnish companies.

SUMMARY:
The study investigates the associations of ambulatory electrodermal activity (EDA) measurements with mental well-being at work, especially job burnout. Appropriate statistical methods are applied to predict burnout with EDA measurements combined with self-report surveys on emotional valence.

DETAILED DESCRIPTION:
The aim of the study is to complement burnout research by considering ambulatory electrodermal activity (EDA) measurements as part of the identification and definition of the burnout phenomenon. Previous studies have shown that assessment methods for the physiological identification of burnout do not yet exist and that more information on the physiological markers of burnout is needed. The study also complements the understanding of how and in what cases ambulatory measurements of EDA can be justified, for example, as an occupational health care tool.

The study investigates the association between ambulatory EDA measurements and mental well-being, especially job burnout, and the potential of the measurements in supporting better mental health at work. According to research the EDA measurements alone do not always provide sufficient information and often context related information is needed to improve the interpretation of the measurement. Therefore, the EDA measurements are complemented with the self-reported emotional valence.

The state of mental well-being is defined using Peter Warr's model of affective well-being. The model proposes that two dimensions of emotion, arousal and emotional valence, together can provide information / be used to describe one's affective well-being at work. The model is further based on the circumplex model of affect.

Previous studies of EDA have shown that the measurement method has a potential role in assisting the diagnosis of some mental disorders, such as anxiety and depression. However, the measurements have been largely tied to laboratory settings and have not been able to be utilized in everyday life. The development of health and well-being technology has brought to the market methods for measuring the electrical conductivity of the skin, which are suitable for ambulatory measurements, but whose suitability must be critically assessed.

Within this study it is hypothesized that the average variation of the sympathetic nervous system activity measured with EDA and combined with a self-reported emotional valence is associated with mental well-being at work, as burnout measured with the Burnout Assessment Tool (BAT-12), anxiety measured with Generalized Anxiety Disorder (GAD-7) Scale, depression measured with Beck Depression Inventory (BDI-21), and job engagement measured with Utrecht Work Engagement Scale (UWES-9).

The study is longitudinal, consisting of four measurement periods at six-month interval. One measurement period of EDA and valence is two weeks. EDA and emotional valence are recorded with a commercially available Moodmetric smart ring and Moodmetric mobile app. EDA is measured with using the Moodmetric index which is calculated from the EDA raw signal produced by the Moodmetric smart ring. EDA and valence measurements are then compared with BAT-12, GAD-7, BDI-21, UWES-9 that measure burnout, anxiety, depression, and job engagement respectively. The survey data (BAT-12, GAD-7, BDI-21, and UWES-9) is gathered after every two-week measurement period is over. 150 voluntary knowledge workers from three Finnish companies are invited to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, but they may have mental health issues
* Employed by one of the target organizations in the beginning of the study
* Informed consent in a written form by the study subject

Exclusion Criteria:

* Nickel sensitivity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Knowledge workers from three Finnish companies.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between electrodermal activity and valence measurements with burnout | Two-weeks
  Association between combined EDA and emotional valence measurements with burnout as measured with BAT-12. The cut-off scores for mild, moderate, and severe burnout are 1.00-2.58, 2.59-3.01 and 3.02-5.00 respectively.

SECONDARY OUTCOMES:
Association between electrodermal activity and valence measurements with anxiety | Two-weeks
  Association between combined EDA and emotional valence measurements with anxiety as measured with GAD-7. The cut-off scores for mild, moderate, and severe anxiety are 5-9, 10-14, 15-21 respectively.
Association between electrodermal activity and valence measurements with depression | Two-weeks
  Association between combined EDA and emotional valence measurements with depression as measured with BDI-21. The cut-off scores for mild mood disturbance, borderline clinical depression, moderate depression, severe depression, and extreme depression are 11-16, 17-20, 21-30, 31-40, and over 40 respectively.
Association between electrodermal activity and valence measurements with job engagement | Two-weeks
  Association between combined EDA and emotional valence measurements with job engagement as measured with UWES-9. Norm scores for very low, low, average, high, and very high are 1.77 or below, 1.78-2.88, 2.89-4.66, 4.67-5.50, and over 5.51 respectively.
Association between electrodermal activity and valence measurements with burnout | Throughout the study 1.5 years: baseline, 6 months, 12 months, and 18 months
  Association between combined EDA and emotional valence measurements with burnout as measured with BAT-12. The cut-off values for mild, moderate, and severe burnout are 1.00-2.58, 2.59-3.01 and 3.02-5.00 respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Saija Mauno, Professor, Study Director — Tampere University
Locations (3):
- Finland (3):
  - Heltti Oy, Helsinki
  - Solita Oy, Helsinki
  - Vincit Oyj, Tampere

IPD SHARING:
Plan to Share IPD: Yes
The following physiological and survey data will be available to other researchers after the study is over, reported and the data irrevocably anonymized:
  * Electrodermal activity measurements recorded with the Moodmetric smart ring
  * Self-reported emotional valence recorded with the Moodmetric mobile app
  * Burnout Assessment Tool (BAT) survey results
  * Beck Depression Inventory (BD1-21) survey results
  * Generalized Anxiety Disorder Scale (GAD-7) survey results
  * Utrecht Work Engagement Scale (UWES-9) survey results
  * Job satisfaction survey results
  The final IPD sharing plan will be made with the assistance of Finnish Social Science Data Archive.
Time Frame: To be determined.
Access Criteria: To be determined.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-04-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT05317793/SAP_000.pdf